CLINICAL TRIAL: NCT07247253
Title: Intervention Efficacy of Assistive Listening Devices for Chinese Children With Dyslexia - a Randomized Controlled Trial
Brief Title: Intervention Efficacy of ALD for Children With Dyslexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, KAM Chi Shan Anna, Associate Professor, Education University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 14150431
Record Dates: First submitted 2025-07-15; First posted 2025-11-25 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Dyslexia
Keywords: Dyslexia; Assistive listening devices; RCT; Chinese
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real ALD (Experimental): Real ALD arm used real ALD (assistive listening device)
  Interventions: Device: Use of a real assistive listening device (FM system) in class.
- Sham ALD (Sham Comparator): Sham ALD arm uses sham ALD (assistive listening device)
  Interventions: Device: Use of a Sham assistive listening device (FM system)

INTERVENTIONS:
Device: Use of a real assistive listening device (FM system) in class. — The Real ALD arm used the real FM system in class.
  Arms: Real ALD
Device: Use of a Sham assistive listening device (FM system) — Use the Sham FM system in class for one year.
  Arms: Sham ALD

SUMMARY:
This double-blind, randomized controlled crossover trial aimed to evaluate the efficacy of providing assistive listening devices (ALDs) in improving specific abilities among Chinese children diagnosed with dyslexia. The primary purpose was to determine whether using ALDs in the classroom setting over the course of one academic year (10 months) leads to significant improvements in literacy abilities compared to using sham (placebo) devices. The study specifically sought to answer the question: Does intervention with real ALDs, as opposed to sham devices, result in superior gains in literacy skills, measured by the change from baseline to 10 months post-intervention initiation? Furthermore, the trial investigated potential treatment benefits on several secondary outcomes, including the neural representation of speech (specifically the consistency of auditory brainstem response to speech sounds), auditory processing abilities, speech and language abilities, phonological awareness, and teachers' perceptions of the children's listening performance in class. The core objective was thus to assess the therapeutic impact of ALDs on literacy development and related auditory and neural functions in this pediatric dyslexic population within their educational environment.

ELIGIBILITY:
Inclusion Criteria:

* aged seven to eleven years;
* diagnosed with dyslexia;
* registered normal IQs (scores > 85);
* displayed normal hearing, with air-conduction thresholds of smaller than or at 25 dB hearing level (HL) for pure tones at octave intervals from 250 Hz to 8000 Hz, with an air-bone gap of < 10 dB for pure tones ranging from 500 Hz to 4000 Hz;
* have not reported current or prior neurological disorders;
* have obtained written informed consent;
* committed to completing the entire study; and
* Chinese who speak Cantonese as the first language.

Exclusion Criteria:

* with known neurological disorders
* with hearing loss
* have not provided written informed consent
* non native Cantonese speaker

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Phonological and orthographic processing - wording reading ability | At enrollment, 10-months after the use of first intervention (real or sham FM system), and 10-months after the use of intervention (sham or real FM system).
  Word reading ability was assessed by counting the number of Chinese character being read correctly in a passage in one minute.
Phonological and orthographic processing - rapid automatized naming | At enrollment, 10-months after the use of first intervention (real or sham FM system), and 10-months after the use of intervention (sham or real FM system).
  A page of randomized letters was presented. The child was required to read the letters row by row as quickly as possible. The number of correctly named letters was counted in one minute.
Orthographic knowledge | At enrollment, 10-months after the use of first intervention (real or sham FM system), and 10-months after the use of intervention (sham or real FM system).
  Orthographic knowledge was assessed by distinguishing real words from nonwords in 20 trials. Percent correct was marked.
Grammar knowledge | At enrollment, 10-months after the use of first intervention (real or sham FM system), and 10-months after the use of intervention (sham or real FM system).
  Grammar knowledge was measured by a sentence reconstruction task. There were 20 items, and the percent correct was marked.
Morphological awareness | At enrollment, 10-months after the use of first intervention (real or sham FM system), and 10-months after the use of intervention (sham or real FM system).
  Morphological awareness was assessed by a homophone identification task. The percent correct on 20 test items was marked.
Reading comprehension | At enrollment, 10-months after the use of first intervention (real or sham FM system), and 10-months after the use of intervention (sham or real FM system).
  A short passage was presented to the kid. The kid was required to answer ten questions based on the understanding of the passage. The percent correct was marked.
Consistency of ABR to sound | At enrollment, 10-months after the use of first intervention (real or sham FM system), and 10-months after the use of intervention (sham or real FM system).
  Consistency of ABR to sound was assessed with this test:
  - An electrophysiological recording protocol that has been employed reliably in previous studies was adopted.16 In brief, the stimuli consisted of 170 ms /ba/, /da/, and /ga/ syllables synthesized with a 50 ms formant transition. In this transition, the first, second, and third formants were dynamic; the fundamental frequency, fourth formant, and fifth formant were stable throughout the process. The stimuli were presented at 80 dB SPL to the right ear monaurally via insert earphones. The polarities of the stimuli alternate at a rate of 4.35 Hz. ABR was captured using a vertical Ag-AgCI electrode montage (Cz active, forehead ground, ipsilateral earlobe reference) in combination with the SmartEP (Intelligence Hearing Systems). A bandpass filter of 70 Hz to 2000 Hz was employed, and a total of 6,000 artifact-free responses (3,000 for each polarity) were obtained for each of the three sounds. Responses from even-numbered events thro

SECONDARY OUTCOMES:
Tone perception ability | At enrollment, 10-months after the use of first intervention (real or sham FM system), and 10-months after the use of intervention (sham or real FM system).
  Tone perception ability was assessed with the Hong Kong Cantonese Tone Identification Test (CANTIT)17.
  - The test consisted of a computerized picture-pointing task. After the target word has been presented auditorily, the subject must select an answer among four choices.
Speech-perception-in-noise ability | At enrollment, 10-months after the use of first intervention (real or sham FM system), and 10-months after the use of intervention (sham or real FM system).
  Speech-perception-in-noise ability was assessed with the Cantonese Hearing in Noise Test (CHINT)18.
  - The test was software-driven and the assessor judged and input the subject's correct or incorrect response for each trial. During the test, speech spectral noise was presented at 70 dB SPL at zero degree azimuth. The presentation level of the target sentence was presented in an adaptive manner (i.e., the presentation of the next target sentence would be decreased by 2 dB for a correct repetition of the current target sentence and vice versa).
Oral language ability | At enrollment, 10-months after the use of first intervention (real or sham FM system), and 10-months after the use of intervention (sham or real FM system).
  Language ability was assessed with the Hong Kong Cantonese Oral Language Assessment Scale (HKCOLAS).
  * HKCOLAS consisted of six subscales: Hong Kong Cantonese grammar, textual comprehension, word definition, lexical-semantic relations, narrative, and expressive nominal vocabulary.
  * The score of each subscale ranges from 1 to 19. The higher the score, the better the performance.
Articulation | At enrollment, 10-months after the use of first intervention (real or sham FM system), and 10-months after the use of intervention (sham or real FM system).
  Articulation was assessed with the Hong Kong Cantonese Articulation test (HKCAT)20.
  - HKCAT consisted of four subscales: consonants, vowels, codas, and tone. The subjects were required to name some pictures.
Phonological awareness | At enrollment, 10-months after the use of first intervention (real or sham FM system), and 10-months after the use of intervention (sham or real FM system).
  Phonological awareness was assessed with a combined test of phoneme rhyme production and phoneme onset deletion.

CONTACTS AND LOCATIONS:
Locations (1):
- The Education University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No